CLINICAL TRIAL: NCT07331220
Title: Pulmonary Artery Denervation for Heart Failure With Preserved Left Ventricular Ejection Fraction
Acronym: PADN-HFpEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Principal Investigator, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20250425-06
Record Dates: First submitted 2025-12-08; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Pulmonary artery denervation; Heart failure with preserved ejection fraction; Guideline-directed medical therapy; Clinical worsening

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to undergo either PADN plus GDMT or sham procedure plus GDMT
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Staff from the core laboratories
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PADN plus GDMT (Experimental): Pulmonary artery denervation combined with guideline-directed medical therapy.
  Interventions: Procedure: PADN; Drug: GDMT
- Sham procedure plus GDMT (Placebo Comparator): Sham procedure combined with guideline-directed medical therapy
  Interventions: Procedure: Sham procedure; Drug: GDMT

INTERVENTIONS:
Procedure: PADN — Advancing the pulmonary artery denervation catheter with a diameter to vessel of 1.1~1.2:1 through the long sheath to the left pulmonary artery ostium. Connecting the catheter to the RF generator. Rotate the catheter under imaging so the premounted electrodes tightly contact the target ablation positions. Recommended temperature-controlled mode, set temperature to 50°C, ablation time to 150 seconds (with effective ablation time of 120 seconds, defined as the tissue temperature reaches 45°C-55°C. Ablation is performed at a total of 3 sites with 120 seconds for each.
  Other Names: Pulmonary artery denervation; Right heart catheterization
  Arms: PADN plus GDMT
Procedure: Sham procedure — The ablation catheter under imaging guidance will be advanced to the target ablation points, but DO NOT connect the ablation catheter to the RF generator; DO NOT deliver RF energy. The operator issues commands to "start" and "stop" RF ablation, simulating the sound of the PADN RF generator for at least 2 minutes (using a pre-recorded MP4).
  Arms: Sham procedure plus GDMT
Drug: GDMT — GDMT regimen including sodium-glucose co-transporter 2 inhibitor (SGLT2i) + spironolactone. SGLT2i can be dapagliflozin or empagliflozin.
  * Dapagliflozin: Target maintenance dose 10 mg/day. Contraindicated if eGFR persistently <25 mL/min/1.73 m².
  * Empagliflozin: Target maintenance dose 10 mg/day. Contraindicated if eGFR persistently <20 mL/min/1.73 m².
  * Spironolactone: Starting dose 10-20 mg/day, maximum dose 40 mg/day. Suspend if serum potassium is >5.5 mmol/L; restart at half dose after correction. Permanently discontinue if serum potassium is >6.0 mmol/L. Suspend and evaluate if eGFR persistently declines >30% or <30 mL/min/1.73 m².
  Other medications are left at the physician's discretion.
  Other Names: Guideline-directed medical therapy

SUMMARY:
To assess the impact of PADN combined with guideline-directed medical therapy (GDMT) versus a sham procedure with GDMT on clinical outcomes in heart failure (HF) patients with preserved left ventricular ejection fraction (LVEF>40%). Outcomes include cardiovascular death, HF-related rehospitalization, requirement for heart transplantation or need of valvular treatment or LVAD or pacemaker implantation, and worsening in outpatients (defined as requirement for intravenous therapy or diuretic intensification, including increasing the types or dose of diuretics).

DETAILED DESCRIPTION:
A randomized, multicenter, blinded, sham-controlled trial in

Subjects with chronic HFpEF (LVEF >40%) meeting inclusion criteria and no exclusion criterion will be enrolled from 25 + centers in China within 24 months. Patients will be randomized 1:1 to:

* Experimental Group: PADN + GDMT
* Control Group: Sham procedure + GDMT

GDMT regimen: Sodium-glucose co-transporter 2 inhibitor (SGLT2i) + Spironolactone. SGLT2i can be dapagliflozin or empagliflozin.

* Dapagliflozin: Target maintenance dose 10 mg/day. Contraindicated if eGFR persistently <25 mL/min/1.73 m².
* Empagliflozin: Target maintenance dose 10 mg/day. Contraindicated if eGFR persistently <20 mL/min/1.73 m².
* Spironolactone: Starting dose 10-20 mg/day, maximum dose 40 mg/day. Suspend if serum potassium is >5.5 mmol/L; restart at half dose after correction. Permanently discontinue if serum potassium is >6.0 mmol/L. Suspend and evaluate if eGFR persistently declines >30% or <30 mL/min/1.73 m².

Other medications are left at the physician's discretion. The proportion of patients with persistent atrial fibrillation is not to exceed 35%.

ELIGIBILITY:
Inclusion Criteria:

1. The subject, or their legal guardian, must have a clear understanding of the trial's design and treatment procedures. They must provide written informed consent before any trial-specific tests or procedures are conducted.

2. Both male and female subjects age between 18 ~ 85 years old. 3. Dyspnea on exertion (NYHA functional class II-IV) not explained by non-cardiac or ischemic etiology.

4. LVEF >40% on imaging within 24 months prior to enrollment, with no clinical changes suggesting worsening systolic function.

5. Elevated NT-proBNP or BNP levels meeting the following thresholds stratified by age and atrial fibrillation (AF) status:

1. Patients WITHOUT atrial fibrillation:

   1. Age <50 years: BNP >100 pg/mL or NT-proBNP >450 pg/mL
   2. Age 50-75 years: BNP >150 pg/mL or NT-proBNP >900 pg/mL
   3. Age >75 years: BNP >200 pg/mL or NT-proBNP >1800 pg/mL
2. Patients WITH atrial fibrillation:

   1. BNP >150 pg/mL or NT-proBNP >300 pg/mL

      6. Stable HF GDMT (no change in either types or dose) for ≥14 days prior to enrollment, including SGLT2i and spironolactone. Other medication, including angiotensin-converting enzyme inhibitors (ACEIs), angiotensin II receptor blockers (ARBs), angiotensin receptor-neprilysin inhibitor (ARNI, sacubitril/valsartan), beta-blockers, or calcium channel blockers (CCBs), were left at physician's discretion.

      7. Dose changes of ACEIs, ARBs, sacubitril/valsartan, beta-blockers, or CCBs did not exceed 100% of baseline dose (i.e., no doubling or halving).

      8. Continuous diuretic use for ≥14 days prior to screening, with stable dose in the last 7 days.

      9. Meet at least one of the following:

   <!-- -->

   1. Hospitalization for decompensated HF within the past 12 months
   2. Received intravenous loop diuretic or ultrafiltration for HF within the past 12 months
   3. Documented resting pulmonary capillary wedge pressure (PCWP) or left ventricular end-diastolic pressure (LVEDP) >15 mmHg, or exercise PCWP ≥25 mmHg, or exercise LVEDP ≥20 mmHg on right heart catheterization within the past 12 months
   4. Echocardiographic evidence within the past 24 months of left atrial enlargement (LA anterior-posterior diameter male >40 mm, female >38 mm; LA area ≥20 cm², LA volume index ≥29 ml/m²) or left ventricular hypertrophy (interventricular septal thickness or LV posterior wall thickness ≥12 mm).

Exclusion Criteria:

1. Hospitalization for HF within 7 days prior to screening.
2. Participation in an interventional trial (using investigational drug or device) of a non-observational registry study within 14 days prior to screening.
3. History of blood or bone marrow donation within 4 weeks prior to screening, or planned donation during the study.
4. Implantation of pulmonary artery pressure monitor or pacemaker within 4 weeks prior to screening, or planned implantation during the study.
5. Hospitalization within 30 days prior to screening for: acute ST-elevation myocardial infarction (STEMI), non-ST-elevation myocardial infarction (NSTEMI), unstable angina, percutaneous coronary intervention (PCI), or cardiac surgery.
6. Cardiac resynchronization therapy (CRT) within 90 days prior to screening.
7. Planned revascularization (PCI or CABG), major cardiac surgery (including coronary artery bypass grafting, valve replacement, ventricular assist device implantation, heart transplantation, other surgery requiring thoracotomy), transcatheter aortic valve replacement (TAVR), or CRT implantation within 90 days after screening.
8. History of femoral or jugular vein surgery.
9. Life expectancy <1 year at screening.
10. Estimated glomerular filtration rate (eGFR) <20 ml/min/1.73 m² at screening (calculated using the modified MDRD formula).
11. BNP <150 pg/ml and NT-proBNP <300 pg/ml at screening.
12. Serum potassium >5.5 mmol/L at screening.
13. Physical examination showing volume depletion at screening or randomization.
14. Mean supine systolic blood pressure <100 mmHg at screening or randomization.
15. Uncontrolled hypertension, defined as mean supine systolic blood pressure ≥160 mmHg (average of three measurements) at screening.
16. Documented stable-state LVEF <40% within the past 24 months.
17. Current active malignancy (excluding non-melanoma skin cancer).
18. HF due to specific cardiomyopathies, including: restrictive/infiltrative cardiomyopathy, active myocarditis, constrictive pericarditis, severe valvular stenosis, hypertrophic obstructive cardiomyopathy (HOCM).
19. Chronic obstructive pulmonary disease (COPD) judged as the primary cause of dyspnea.
20. Myocardial ischemia judged as the primary cause of dyspnea.
21. Isolated right heart failure due to pulmonary disease.
22. Complex congenital heart disease.
23. History of allergic reaction to guideline-directed HF medications.
24. Pregnant/lactating women. Women of childbearing potential (WOCBP) defined as post-menarche and not permanently sterilized (hysterectomy/bilateral tubal ligation) or postmenopausal (natural amenorrhea ≥12 months without other medical cause). Sexually active WOCBP must agree to use medically accepted contraception during the study, including: |surgical sterilization, progestin contraceptives (oral/implant), barrier methods (condom/diaphragm) with spermicide, intrauterine device (IUD). Urine pregnancy test required at each visit; negative result required for continued participation.
25. Other exclusion criteria as judged by the investigator, including but not limited to conditions that may jeopardize patient safety during study participation, factors interfering with study data interpretation, or patients unlikely to comply with study procedures/requirements.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical worsening | From randomization to 12 months
  A composite of clinical worsening at 12 months, including cardiovascular death, HF-related rehospitalization, requirement for heart transplantation, need of valvular treatment or LVAD or pacemaker implantation, and worsening in outpatients (defined as requirement for intravenous therapy or diuretic intensification, including increasing the types or dose of diuretics).

SECONDARY OUTCOMES:
Clinical worsening | From baseline to 24 months
  A composite of clinical worsening at 24 months, including cardiovascular death, HF-related rehospitalization, requirement for heart transplantation, need of valvular treatment or LVAD or pacemaker implantation, and worsening in outpatients (defined as requirement for intravenous therapy or diuretic intensification, including increasing the types or dose of diuretics).
Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS) | From baseline to 12 months
  The Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS) is a percentage-based health index ranging from 0 to 100, where higher scores indicate better heart failure-related health status.
N-terminal pro-B-type natriuretic peptide (NT-proBNP) | From baseline to 1 month, 6 months, and 12 months
  Change in NT-proBNP levels at 1 month, 6 months, and 12 months.
6-minute walk distance (6MWD) | From baseline to 1 month, 6 months, and 12 months
  The 6-minute walk test in patients with chronic heart failure is clinically graded as follows: A distance of less than 150 meters indicates severe heart failure with poor prognosis; 150 to 300 meters corresponds to moderate heart failure; 300 to 450 meters reflects mild heart failure; and a distance greater than 450 meters suggests near-normal cardiac function and a relatively better clinical status.
KCCQ-CSS increase ≥6 points | From baseline to 12 months
  The Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS) is a percentage-based health index ranging from 0 to 100, where higher scores indicate better heart failure-related health status.
NT-proBNP reduction ≥20% | From baseline to 6 months and 12 months
  Proportion of patients with NT-proBNP reduction ≥20% at 6, 12 months
KCCQ-CSS increase ≥6 points and NT-proBNP reduction ≥20% | From baseline to 6 months and 12 months
  KCCQ-CSS and NT-proBNP will be combined to report heart failure-related health status.
Echocardiographic parameters (chamber size, systolic and diastolic function) | From baseline to 6 months
  Echocardiographic parameters, such as left ventricular ejection fraction (LVEF), ventricular volumes, and diastolic function indices (e.g., E/e' ratio), serve as key quantitative endpoints to evaluate cardiac remodeling and therapeutic response.
Rate of worsening in outpatients | Within 12 months
  requiring intravenous injection of medicines, or needing diuretic intensification (including increase in types or doses of diuretics).
Rate of heart or lung transplantation | within 12 months
  For patients with progressive heart failure
Rate of left ventricular assist device implantation | Within 12 months
  Incidence of left ventricular assist device (LVAD) implantation, defined as the proportion of patients undergoing LVAD surgery during the study follow-up period.
Requirement of pacemaker / physiologic pacing / CRT / ICD/valvular treatment | Within 12 months
  Indications for pacemaker: Symptomatic sinus node dysfunction, High-grade AV block (Mobitz II or complete heart block), and Post-TAVI or post-MI advanced conduction disease when persistent.
  Indications for CRT: LVEF ≤35%, Sinus rhythm, LBBB morphology, QRS ≥150 ms, NYHA II-III or ambulatory IV, or others (determined by EP team).
  Indications for valvular treatment: Aortic Stenosis (AS), Aortic Regurgitation (AR) with Symptoms or Asymptomatic but LVEF ≤55% and/or progressive LV dilation, Primary (degenerative) Mitral Regurgitation (MR) Symptoms or LV dysfunction developing (LVEF ≤60%, Tricuspid Regurgitation (TR), Mitral Stenosis (MS), or others.
All events within 24 months | Within 24 months
  All patients will be followed-up until 24 months

OTHER OUTCOMES:
Loop diuretic dose | From baseline to 12 months
  Weekly loop diuretic dose (furosemide equivalent) change
SGLT2i dose | From baseline to 12 months
  Weekly SGLT2i dose (dapagliflozin or empagliflozin) change
NYHA functional class | From baseline to 12 months
  Change in New York Heart Association (NYHA) functional class at 12 months.
Mortality | From baseline to 12 months
  All-cause mortality
Cardiovascular mortality | From baseline to 12 months
Rate of non-fatal myocardial infarction | From baseline to 12 months
Rate of stroke | From baseline to 12 months
Rate of acute kidney injury | From baseline to 12 months
  Acute kidney injury (serum creatinine doubling based on modified RIFLE criteria).
Adverse events (AEs) and Serious Adverse Events (SAEs) | From baseline to 12 months
  Adverse events (AEs) and Serious Adverse Events (SAEs), including access site complications (e.g., bleeding, hematoma).

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
DATA sharing could be accepted upon other researchers reached out to the PI of this trial, with approval.
Supporting Information: Analytic Code
Time Frame: It will be available after 6 months since publication of this trial, unless PI agreed earlier.
Access Criteria: upon approval by PI of this trial